CLINICAL TRIAL: NCT04863027
Title: PHASE I-II Study on the Use of Dual Energy Computed Tomography for Assessment of Lung Function in Thoracic Conventional and Stereotactic Body Radiotherapy
Brief Title: Use of Dual Energy Computed Tomography in Thoracic Radiotherapy Planning.
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: 14.003
Record Dates: First submitted 2021-03-29; First posted 2021-04-28 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Lung Cancer; Lung Function Decreased; Radiation Pneumonitis
MeSH Terms: conditions — Lung Neoplasms; Respiratory Insufficiency; Radiation Pneumonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Thoracic radiotherapy — Patients will have pre-treatment and post-treatment perfusion DECT for baseline and post-treatment lung function

SUMMARY:
This is a prospective observational study aiming: 1) To quantify lung function using perfusion dual energy computed tomography (DECT) and use this information at the time of treatment planning with preferential sparing of functional lung parenchymal 2) to validate results of lung function obtained using DECT with lung perfusion scintigraphy results, the current standard method; 4) to compare dosimetry of whole lungs vs. functional lungs in patients treated with either stereotactic body radiotherapy (SBRT) for early stage lung cancer or conventional radiotherapy for locally advanced lung cancer and 5) to evaluate lung function 6, 12 and 24 months post-radiotherapy with both perfusion DECT and pulmonary function tests and compare radiation dose-map to functional lung-map.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* ECOG 0-2
* Pulmonary neoplasia, confirmed histopathologically or by imaging
* Prognosis evaluated ≥ 1 year by attending MD
* Clinically acceptable lung capacity to undergo radiotherapy
* Initial assessment including history, physical examination, biochemistry, PFT, chest radiograph, chest and abdominal-pelvic scan, PET
* Written consent
* The patient must be available for treatment and monitoring. Patients registered in the study should be treated in our center.

Exclusion criteria

* Previous radiotherapy in the radiation field
* Presence of any major medical condition that, in the opinion of the investigator, would prevent follow-up at 6, 12 and 24 months post-radiotherapy.
* Iodine allergy
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer planned for curative intent radiotherapy (conventional or stereotactic)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Lung function quantification at baseline | Baseline
  To quantify lung function using perfusion DECT and use this information at the time of treatment planning with preferential sparing of functional lung parenchyma.
Radiation-induced lung function damage quantification | at 12 months after radiotherapy
  To evaluate lung function post-radiotherapy with both perfusion DECT and pulmonary function tests and compare radiation dose-map to functional lung-map.
Radiation-induced lung function damage quantification | at 24 months after radiotherapy
  To evaluate lung function post-radiotherapy with both perfusion DECT and pulmonary function tests and compare radiation dose-map to functional lung-map.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided